CLINICAL TRIAL: NCT02356991
Title: A Randomized,Double-Blind, Placebo-Controlled, Multicenter, Phase II Study of Famitinib in Patients With Advanced Non-squamous and Non-Small Cell Lung Cancer (NSCLC)
Brief Title: A Study of Famitinib in Patients With Advanced Non-squamous and Non-Small Cell Lung Cancer (NSCLC)
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: sponsor decides to suspend this trial
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Collaborators: Sun Yat-sen University (Other); Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HR-FMTN- Ⅱ-NSCLC-MON
Record Dates: First submitted 2015-01-16; First posted 2015-02-06 (Estimated); Last update posted 2019-11-04 (Actual); Status verified 2019-10

CONDITIONS: Non-Small Cell Lung Cancer (NSCLC)
Keywords: Famitinib; Phase II; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — famitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Famitinib (Experimental): Famitinib 25 mg qd p.o., 4 weeks per cycle.The treatment continued until disease progression or intolerable toxicity happened or patients withdrawal of consent.
  Interventions: Drug: Famitinib
- Placebo (Placebo Comparator): Placebo 25 mg qd p.o., 4 weeks per cycle.The treatment continued until disease progression or intolerable toxicity happened or patients withdrawal of consent.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Famitinib
  Arms: Famitinib
Drug: Placebo
  Arms: Placebo

SUMMARY:
Famitinib is a tyrosin-inhibitor agent targeting at c-Kit, VEGFR2, PDGFR, VEGFR3, Flt1 and Flt3. Phase I study has shown that the toxicity is manageable.

The purpose of this study is to evaluate the efficacy and safety profile of Famitinib in patients with Advanced Non-squamous and Non-Small Cell Lung Cancer (NSCLC).

ELIGIBILITY:
Inclusion Criteria:

* 1.Age: 18-70;
* 2.Advanced (IV phase)non squamous NSCLC confirmed by pathology, with measurable lesions (tumour lesions ≥10mm in longest diameter, malignant lymph nodes ≥15mm in short axis, scanning layer ≤ 5 mm, measurable lesions not received locoregional theraphy ,such as radiotherapy or frozen therapy);
* 3.Previously treated with EGFR inhibitors or chemotherapy,second line or above treatment failure:

  * a.for EGFR wild type, second line or above treatment failure(at least previously treated with platinum-based chemotherapy)
  * b.for EGFR mutation type, third line or above treatment failure(at least previously treated with Platinum-based chemotherapy and EGFR inhibitors)
* 4.ECOG Performance Status of 0 or 1;
* 5.Life expectancy of at least 3 months;
* 6.Damage caused by other anti-tumor therapy has been restored, the nitroso or mitomycin treatment interval ≥ 6 weeks; other cytotoxic drugs, radiotherapy or surgery for ≥ 4 weeks; EGFR molecular targeted drugs for ≥ 2 weeks;
* 7.Participants have inadequate organ and marrow function as defined below:

  * Hemoglobin ≥ 90g/L ( no blood transfusion in 2 weeks)
  * Absolute neutrophil count (ANC) ≥ 1.5×10^9/L
  * PLT ≥ 80×10^9/L
  * Bilirubin < 1.25 × ULN
  * ALT < 2.5 × ULN
  * AST < 2.5 × ULN
  * serum creatinine < 1.25 × ULN, and endogenous Cr clearance > 45 ml/min(Cockcroft-Gault Formula)
  * cholesterol ≤ 1.5×ULN and triglyceride≤ 2.5 × ULN
  * LVEF≥ LLN by Color Doppler Ultrasonography
* 8.Female: Child bearing potential, a negative urine or serum pregnancy test result 7 days before initiating famitinib.All subjects who are not surgically sterile or postmenopausal must agree and commit to the use of a reliable method of birth control for the duration of the study and for 8 weeks after the last dose of test article. Male: All subjects who are not surgically sterile or postmenopausal must agree and commit to the use of a reliable method of birth control for the duration of the study and for 8 weeks after the last dose of test article;
* 9.Ability to understand and willingness to sign a written informed consent. Good compliance with follow-up visits.

Exclusion Criteria:

* 1.Squamous cell carcinoma (including adenosquamous carcinoma, undifferentiated carcinoma); small cell lung cancer (lung cancer including small cell carcinoma and non-small cell hybrid);
* 2.Known brain metastases, spinal cord compression, cancer meningitis, or screening CT or MRI examination revealed brain or leptomeningeal disease
* 3.Patients with hypertension using combination therapy (systolic blood pressure> 140 mmHg, diastolic blood pressure> 90 mmHg). Patients with more than Class I, myocardial ischemia or myocardial infarction, arrhythmia (including QT interval ≥ 450ms for male and 470ms for female) and class II cardiac dysfunction,according to NCI-CTC AE 4.0;
* 4.Variety of factors that affect the oral medication (such as inability to swallow, gastrointestinal resection, chronic diarrhea and intestinal obstruction);
* 5.Coagulation abnormalities (PT or PT-INR > 1.5 ULN, and APTT > 1.5 ULN), bleeding tendency (eg, active peptic ulcer) or are receiving thrombolytic or anticoagulant therapy;
* 6.Distance between tumours lesions and major blood vessels with radiographical evidence (CT or MRI) ≥5mm.
* 7.Pulmonary hemorrhage/ bleeding event ≥ CTCAE gr. 1 （including Hemoptysis≥2.5ml or half teaspoon）within four weeks of the first dose of the study drug; Any other hemorrhage/ bleeding event ≥ CTCAE gr. 2 within four weeks of the first dose of the study drug;
* 8.Long-term untreated wounds or fractures;
* 9.Thrombotic or embolic venous or arterial events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis or pulmonary embolism within the 12 months prior to the first dose of study drug;
* 10.Urine protein ≥ + + and confirmed the 24-hour urinary protein>1.0 g;
* 11.Application of anticoagulants or vitamin K antagonists such as warfarin, heparin or its analogues; If the prothrombin time international normalized ratio (INR) ≤ 1.5, with the purpose of prevention, the use of small doses of warfarin (1mg orally, once daily) ，low-dose heparin (0.6~1.2 ×10^8 U daily) low-dose aspirin (less than 100mg daily) is allowed;
* 12.Preexisting thyroid dysfunction, even using medical therapy, thyroid function cannot maintain in the normal range;
* 13.Pre-existing ascites and/or clinically significant pleural effusion;
* 14.Active hepatitis C and/or B infection;
* 15.Abuse of psychiatric drugs or dysphrenia;
* 16.Participated in other anti-cancer clinical trials within four weeks;
* 17.Prior therapy with VEGFR inhibitor，except Bevacizumab (Avastin);
* 18.Past or suffering from other cancer, but other than cure basal cell carcinoma and cervical carcinoma in situ.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Progress free survival (PFS) | 1.5 years

SECONDARY OUTCOMES:
Overall Survival (OS) | 2 years
Objective Response Rate (ORR) | 1 years
Disease Control Rate (DCR) | 1 years
Quality of Life | 28-day cycle visit until disease progress

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, M.D., Principal Investigator — Cancer Hospital of Guangzhou Sun Yat-sen University
Locations (2):
- China (2):
  - Cancer Hospital of Guangzhou Sun Yat-sen University, Guangzhou, Guangdong
  - Tongji University Affiliated Shanghai Pulmonary Hospital, Shanghai